CLINICAL TRIAL: NCT04624230
Title: OPEN-LABEL INDUCTION AND MAINTENANCE STUDY OF ORAL CP-690,550 (TOFACITINIB) IN CHILDREN WITH MODERATELY TO SEVERELY ACTIVE ULCERATIVE COLITIS
Brief Title: Evaluation of Oral Tofacitinib in Children Aged 2 to 17 Years Old Suffering From Moderate to Severe Ulcerative Colitis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: A3921210; OVATION (Other: Alias Study Number); 2023-509694-22-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2020-10-26; First posted 2020-11-10 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Pediatric; Tofacitinib Oral; Mayo; PUCAI; Flare
MeSH Terms: conditions — Colitis, Ulcerative | interventions — tofacitinib

STUDY DESIGN:
Intervention Model Description: Single Group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- tofacitinib (Experimental): Open label tofacitinib 5 mg BID weight based adult equivalent with the option for individual dose increase to 10 mg BID weight based adult equivalent for a limited time if dose escalation criteria are met, prior to returning to 5 mg BID.
  Interventions: Drug: tofacitinib

INTERVENTIONS:
Drug: tofacitinib — Open label tofacitinib 5 mg BID weight based adult equivalent with the option for individual dose increase to 10 mg BID weight based adult equivalent for a limited time if dose escalation criteria are met, prior to returning to 5 mg BID.

SUMMARY:
This study, A3921210 is designed to evaluate the efficacy, safety and pharmacokinetics (PK) of tofacitinib in pediatric participants with moderately to severely active UC. In the US and EU, patients with prior TNFi failure or intolerance will be enrolled. Outside of the US or EU, patients having had inadequate response or intolerance to oral or IV corticosteroids or azathioprine or 6-mercaptopurine or TNFi will be enrolled.

All eligible participants will initially receive open label tofacitinib at a dose expected to produce equivalent systemic exposure to that observed in adults receiving 5 mg BID with the option for individual dose increase to 10 mg BID adult dose equivalent if dose escalation criteria are met.

The primary objective of this study is to evaluate the efficacy of tofacitinib based on remission in pediatric participants with moderately to severely active UC. The primary endpoint is remission by central read Mayo score following 44 weeks in the maintenance phase. Remission is defined by a Mayo score of 2 points or lower, with no individual subscore exceeding 1 point and a rectal bleeding subscore of 0.

The study Design is an open-label Phase 3 study that includes a screening period of up to 4-weeks duration, an 8-week or 16-week induction phase, a 44-week maintenance phase, and a 24-month extension phase for pediatric participants with moderately to severely active UC. Participants will have a follow-up visit 4 weeks after the last dose of study intervention and a telephone contact 8 weeks later to assess for any adverse events (AEs)/serious adverse events (SAEs). The total maximum duration of this study will be up to 180 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document and assent document.
* Males and females 2 to less than18 years old and weighing at least 10 kg.
* Having a pathology report that confirms colonic inflammation consistent with UC with a clinical diagnosis of UC for at least 12 weeks prior to baseline, with biopsy report supporting the diagnosis of UC.
* Participants diagnosed with UC at age less than 6 years old, must have had testing and be negative for monogenic disorders associated with very early onset IBD.
* Moderately to severely active UC as defined (via screening colonoscopy) by a Mayo score of at least 6, with a rectal bleeding score of at least 1 and an endoscopic subscore of at least 2.
* Pediatric Ulcerative Colitis Activity Index (PUCAI) score greater or equal to 35 .
* No history of dysplasia or colon cancer.
* No evidence or history of untreated or inadequately treated active or latent infection with Mycobacterium Tuberculosis.
* For participants outside of the United States or the European Union: have had an inadequate response or been intolerant to at least one prior therapy as listed below or have a medical contraindication to such therapies:

  * Oral or intravenous (IV) corticosteroids;
  * Azathioprine or 6-mercaptopurine;
  * TNF inhibitors or anti integrin therapy.
* For participants in the United States and the European Union: have had an inadequate response or intolerance to TNF inhibitors.
* Stable doses of the following therapies for UC:

  * Oral 5 Aminosalicyclic acids (ASA) or sulfasalazine
  * Oral corticosteroids equivalent to prednisone at most 1 mg/kg up to a maximum of 20 mg/day or budesonide up to 9 mg/day.
* female participant is eligible if she is not pregnant or breastfeeding, If she is a woman of child bearing potential, she needs to be using a contraceptive method that is highly effective (with a failure rate of <1% per year).

Exclusion Criteria:

* Diagnosis of indeterminate colitis, isolated proctitis, microscopic colitis, infectious colitis, Crohn's disease, or clinical findings suggestive of Crohn's disease.
* History of symptomatic obstructive intestinal strictures or active ostomy, or history of colectomy, extensive small bowel resection ( greater than100 centimetres) or short bowel syndrome, or hospitalization for UC related reason(s) within 2 weeks of baseline visit.
* Any factors or clinical characteristics potentially related to the risk of venous thromboembolism that may increase the risk associated with study participation or study intervention administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Participants who have previously received tofacitinib or another Janus Kinase inhibitor.
* Vaccination or exposure to a live or attenuated vaccine within the 6 weeks prior to the first dose of study drug, or who are expected to be vaccinated or to have household exposure to these vaccines during treatment or during the 6 weeks following discontinuation of study drug.
* Participants having received azathioprine, 6-mercaptopurine, methotrexate, thioguanine, infliximab, adalimumab, golimumab, ustekinumab, interferon, cyclosporine, mycophenolate, tacrolimus, IV or rectally administered corticosteroids, natalizumab, vedolizumab, other antiadhesion molecules, or investigational drugs during the specified time periods prior to baseline whereby they may still have pharmacokinetic and/or pharmacodynamic effect in the body of the participant.
* Previous treatment by leukocyte apheresis including selective lymphocyte, monocyte, or granulocyte apheresis, or plasma exchange within 6 months prior to baseline.
* Treatment by specified prohibited concomitant medications, including moderate to potent CYP3A inducers or inhibitors in the specified time periods prior to the first dose of study drug or are expected to receive any of these medications during the study period.
* Chronic and frequent use of antimotility agents for control of diarrhea (ie, diphenoxylate hydrochloride with atropine sulfate or loperamide).
* History of bowel surgery, including cholecystectomy within 6 months prior to baseline, history of appendectomy within 3 months prior to baseline, or significant trauma or major surgery within 4 weeks of screening visit are excluded.
* Participants with the following laboratory values at screening:

  * Hemoglobin level lower than 9.0 g/Dl.
  * Absolute white blood cell (WBC) count lower than 3000/mm3.
  * Absolute neutrophil count lower than 1200/mm3.
  * Absolute lymphocyte count lower than 750/mm3.
  * Thrombocytopenia as defined by a platelet count lower than 100,000/mm3.
  * Estimated bedside Schwartz Glomerular filtration rate (GFR) lower or equal to 40 mL/min/1.73 m2.
  * Total bilirubin, aspartate aminostransferase (AST) or alanine aminotransferase (ALT) more than 1.5 times the upper limit of normal.
* Positive stool examinations for enteric pathogens, pathogenic ova or parasites, or C. difficile toxin at screening.
* Participants infected with human immunodeficiency virus (HIV) or hepatitis B or C viruses.
* History of more than one episode of HZ, a history of disseminated HZ or disseminated herpes simplex.
* History or current symptoms of any lymphoproliferative disorder (eg, Epstein Barr Virus (EBV) related lymphoproliferative disorder, lymphoma, leukemia, myeloproliferative disorders, multiple myeloma, or signs and symptoms suggestive of currently lymphatic disease).
* Clinically significant infections currently or within 3 months prior to baseline (eg, those requiring hospitalization or parenteral antimicrobial therapy or opportunistic infections), a history of any infection requiring antimicrobial therapy within 2 weeks of baseline, or a history of any infection otherwise judged by the investigator to have the potential for exacerbation by participation in the study.
* Any malignancies or with a history of malignancies, with the exception of adequately treated or excised nonmetastatic basal cell or squamous cell cancer of the skin.
* Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or participants who are employees of the Sponsor, including their family members, directly involved in the conduct of the study.
* Participation in other studies involving investigational drug(s) within 2 months prior to study entry and/or during study participation.
* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or study intervention administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Pregnant female participants; breastfeeding female participants; fertile female participants of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and through the telephone follow up visit.
* History of allergies, intolerance or hypersensitivity to lactose or tofacitinib, or any other excipients of the investigational medicinal products, including placebos.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2021-08-12 (Actual); Primary Completion 2027-02-23 (Estimated); Study Completion 2029-05-15 (Estimated)

PRIMARY OUTCOMES:
Remission by central read Mayo score following 44 weeks in the maintenance phase. | Outcome measured at the end of the 44 weeks of the maintenance phase.
  Remission is defined by central endoscopy read Mayo score of 2 points or lower, with no individual subscore exceeding 1 point and a rectal bleeding subscore of 0.
  The primary outcome Mayo score is the summation of 4 subscores as listed below :
  * patient reported stool frequency (scored 0 to 3)
  * patient reported rectal bleeding (scored 0 to 3)
  * central read findings on endoscopy (scored 0 to 3)
  * physician's global assessment (scored 0 to 3)
  The Mayo score has a scale from 0 to 12 points, with the lower score indicating lower ulcerative colitis (UC) disease activity.

SECONDARY OUTCOMES:
Response by Mayo score | Outcome measured at induction Week 8, induction Week 16, and maintenance Week 44
  Response by Mayo score is defined by a decrease from baseline in Mayo score of at least 3 points and at least 30%, with an accompanying decrease in the subscore for rectal bleeding of at least 1 point or absolute subscore for rectal bleeding of 0 or 1.
Remission by Mayo score | Outcome measured at induction Week 8, induction Week 16, and maintenance Week 44
  Remission by Mayo score with local and central endoscopy read (induction Week 8, induction Week 16), and with local endoscopy read only (maintenance week 44).
Change from baseline in Mayo score. | Outcome measured at induction Week 8, induction Week 16, and maintenance Week 44
Response measured by Partial Mayo Score | Outcome measured through study completion, an average of 3 and a half years
  Response is defined by a partial Mayo score decrease of 2 points or more from baseline. This score is based on the summation of the following subscores :
  * stool frequency (scored 0 to 3)
  * rectal bleeding (scored 0 to 3)
  * physician global assessment (PGA) (scored 0 to 3)
  The partial Mayo score has a scale from 0 to 9, with the lower score indicating lower ulcerative colitis (UC) disease activity.
Change from baseline in Partial Mayo score | Outcome measured through study completion, an average of 3 and a half years
  Change in partial Mayo score. This score is the summation of 3 distinct dimensions as listed below :
  * stool frequency (scored 0 to 3)
  * rectal bleeding (scored 0 to 3)
  * physician global assessment (PGA) (scored 0 to 3)
  The partial Mayo score has a scale from 0 to 9, with the lower score indicating lower ulcerative colitis (UC) disease activity.
Response by PUCAI score | Outcome measured through study completion, an average of 3 and a half years
  The Pediatric Ulcerative Colitis Activity Index (PUCAI) score is the summation of 6 dimensions that are all reported by the investigator. The PUCAI score varies from 0 to 85 points, with the lower score indicating lower ulcerative colitis (UC) disease activity. The 6 dimensions of the PUCAI score are as follows :
  * abdominal pain
  * rectal bleeding
  * stool consistency of most stools
  * number of stools per 24 hours
  * nocturnal stools
  * activity level
  Response is defined by a PUCAI score decrease of 20 points or more.
Change from baseline in PUCAI score | Outcome measured through study completion, an average of 3 and a half years
  The Pediatric Ulcerative Colitis Activity Index (PUCAI) score is the summation of 6 dimensions that are all reported by the investigator
  * abdominal pain
  * rectal bleeding
  * stool consistency of most stools
  * number of stools per 24 hours
  * nocturnal stools
  * activity level
  The PUCAI score varies from 0 to 85 points, with the lower score indicating lower ulcerative colitis (UC) disease activity.
Percentage of Participants Achieving Endoscopic Improvement at Week 8, 16, and 44 | Outcome measured at induction Week 8, induction Week 16, and maintenance Week 44
  Endoscopic improvement is defined by Mayo endoscopic sub-score of 0 or 1. The Mayo endoscopic sub-score is used to assess ulcerative colitis activity, and ranges from 0 to 3, and is based on the findings during endoscopy. A lower score is indicative of a lower ulcerative colitis (UC) disease activity.
Time to flare | Outcome measured from 2 to 4 months in the study, through study completion, an average of 3 and a half years
Change from baseline in fecal calprotectin levels | Outcome measured through study completion, an average of 3 and a half years
Change from baseline in serum high sensitivity C-Reactive Protein (hsCRP) levels | Outcome measured through study completion, an average of 3 and a half years
Corticosteroid free remission by Partial Mayo Score | Outcome measured through study completion, an average of 3 and a half years
  Remission is defined by a partial Mayo score of 2 points or lower, with no individual subscore exceeding 1 point and rectal bleeding subscore of 0.
  The subscores of the partial Mayo score are:
  * stool frequency (scored 0 to 3)
  * rectal bleeding (scored 0 to 3)
  * physician global assessment (PGA) (scored 0 to 3)
Average plasma concentration of tofacitinib (Cavg) | Outcome measured at baseline, induction Week 8, induction Week 16, maintenance Week 16, maintenance Week 44
Evaluation of taste acceptability of tofacitinib oral solution, and acceptability of film coated tablet by choosing one of 5 choices | Outcome measured at induction week 2
  Taste acceptability will be assessed by asking the participant to select one of 5 choices which most adequately reflects the participant's response to taste. Age appropriate tools (using wording and/or graphic facial expressions) will be used to assess taste acceptability.
Peak (maximum) plasma concentration of tofacitinib (Cmax) | Outcome measured at baseline, induction Week 8, induction Week 16, maintenance Week 16, maintenance Week 44
Percentage of Participants Achieving Endoscopic Remission at Week 8, 16, and 44 | Outcome measured at induction Week 8, induction Week 16, and maintenance Week 44
  Endoscopic remission is defined by a Mayo endoscopic subscore of 0, out of a maximum of 3 points.
  The Mayo endoscopic sub-score is used to assess ulcerative colitis activity, and ranges from 0 to 3, and is based on the findings during endoscopy. A lower score is indicative of a lower ulcerative colitis (UC) disease activity.
Remission by PUCAI score | Outcome measured through study completion, an average of 3 and a half years
  The Pediatric Ulcerative Colitis Activity Index (PUCAI) score is the summation of 6 dimensions that are all reported by the investigator. The PUCAI score varies from 0 to 85 points, with the lower score indicating lower ulcerative colitis (UC) disease activity. The 6 dimensions of the PUCAI score are as follows :
  * abdominal pain
  * rectal bleeding
  * stool consistency of most stools
  * number of stools per 24 hours
  * nocturnal stools
  * activity level
  Remission is defined by a PUCAI score of less than 10 points.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (77):
- United States (24):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California, San Francisco Benioff Children's Hospital, San Francisco, California
  - University of California, San Francisco Pediatric Clinical Research Center (PCRC), San Francisco, California
  - Connecticut Children's Ambulatory Surgical Center, Farmington, Connecticut
  - Connecticut Children's Infusion Center, Farmington, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Nicklaus Children's Hospital, Miami, Florida
  - Center for Advanced Pediatrics, Atlanta, Georgia
  - Children's Healthcare of Atlanta - Arthur M. Blank Hospital, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - Atlantic Children's Health-Pediatric Gastroenterology & Nutrition, Morristown, New Jersey
  - Goryeb Children's Hospital (Endoscopy only), Morristown, New Jersey
  - Atlantic Health System- Morristown Medical Center (Pharmacy), Morristown, New Jersey
  - Northwell Health - Cohen Children's Medical Center, Lake Success, New York
  - Northwell Health - Cohen Children's Medical Center, New Hyde Park, New York
  - Columbia University Irving Medical Center, New York, New York
  - CUIMC Research Pharmacy - Milstein Hospital (Pharmacy Only), New York, New York
  - Morgan Stanley Children's Hospital, CUIMC, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Buerger Center for Advanced Pediatric Care, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Roberts Center for Pediatric Research, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- The Royal Children's Hospital, Parkville, Victoria, Australia
- Belgium (4):
  - Universitaire Ziekenhuizen Leuven, Leuven, Vlaams Brabant
  - Hôpital Universitaire Des Enfants Reine Fabiola, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
- Canada (6):
  - Stollery Children's Hospital University of Alberta, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - London Health Sciences Centre - Children's Hospital, London, Ontario
  - The Hospital for Sick Children - Division of Gastroenterology, Hepatology and Nutrition, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
- Tampereen yliopistollinen sairaala, Tampere, Finland
- France (2):
  - CHU de Lyon - Hôpital Femme Mère Enfant, Bron
  - Hôpital Necker Enfants Malades, Paris
- Dr. von Haunersches Kinderspital, LMU, Munich, Bavaria, Germany
- Hungary (2):
  - Debreceni Egyetem Klinikai Kozpont, Debrecen, Hajdú-Bihar
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
- Israel (5):
  - Shamir Medical Center (Assaf Harofeh), Be’er Ya‘aqov
  - Lady Davis Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Schneider Children's Medical Center of Israel, Petah Tikva
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (4):
  - ASST Papa Giovanni XXIII Epatologia e Gastroenterologia Pediatrica e dei Trapianti, Bergamo, BG
  - A.O.U. Federico II, Napoli, Naples
  - Azienda Ospedaliero - Universitaria Policlinico Umberto I di Roma, Roma, RM
  - Azienda USL di Bologna - IRCCS ISNB - Programma Gastroenterologia Pediatrica, Bologna
- Japan (10):
  - Aichi Children's Health and Medical Center, Obu-shi, Aichi-ken
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Gunma University Hospital, Maebashi, Gunma
  - Miyagi Children's Hospital, Sendai, Miyagi
  - Osaka Women's and Children's Hospital, Izumi, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki-shi, Osaka
  - Saitama Prefectural Children's Medical Center, Saitama-shi, Saitama
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - National Center for Child Health and Development, Setagaya-ku, Tokyo
- Netherlands (3):
  - Amsterdam UMC location AMC, Amsterdam, North Holland
  - Amsterdam UMC, location VUmc Boelelaan, Amsterdam
  - Erasmus Medical Center - Sophia Children's Hospital, Rotterdam
- Poland (5):
  - Medical Network Spółka z o.o. WIP Warsaw IBD Point Profesor Kierkuś, Warsaw, Masovian Voivodeship
  - Instytut "Centrum Zdrowia Matki Polki", Lodz
  - Korczowski Bartosz, Gabinet Lekarski, Rzeszów
  - Instytut "Pomnik - Centrum Zdrowia Dziecka", Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw
- Narodny ustav detskych chorob, Bratislava, Slovakia
- Hospital Infantil Universitario Niño Jesus, Madrid, Spain
- Sweden (3):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Sachsska Children's and Youth Hospital/South General Hospital, Stockholm
  - Karolinska Universitetssjukhuset Barngastroenterologi, hepatologi och nutrition, Stockholm
- United Kingdom (4):
  - King's College Hospital NHS Foundation Trust, London, Greater London
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham, WEST Midlands
  - NHS Lothian, Edinburgh
  - Bart's Health NHS Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Result] Benchimol EI, Bernstein CN, Bitton A, Carroll MW, Singh H, Otley AR, Vutcovici M, El-Matary W, Nguyen GC, Griffiths AM, Mack DR, Jacobson K, Mojaverian N, Tanyingoh D, Cui Y, Nugent ZJ, Coulombe J, Targownik LE, Jones JL, Leddin D, Murthy SK, Kaplan GG. Trends in Epidemiology of Pediatric Inflammatory Bowel Disease in Canada: Distributed Network Analysis of Multiple Population-Based Provincial Health Administrative Databases. Am J Gastroenterol. 2017 Jul;112(7):1120-1134. doi: 10.1038/ajg.2017.97. Epub 2017 Apr 18. PMID 28417994
- [Result] Konstantinides SV, Meyer G, Becattini C, Bueno H, Geersing GJ, Harjola VP, Huisman MV, Humbert M, Jennings CS, Jimenez D, Kucher N, Lang IM, Lankeit M, Lorusso R, Mazzolai L, Meneveau N, Ni Ainle F, Prandoni P, Pruszczyk P, Righini M, Torbicki A, Van Belle E, Zamorano JL; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of acute pulmonary embolism developed in collaboration with the European Respiratory Society (ERS). Eur Heart J. 2020 Jan 21;41(4):543-603. doi: 10.1093/eurheartj/ehz405. No abstract available. PMID 31504429
- [Result] Kelsen JR, Sullivan KE, Rabizadeh S, Singh N, Snapper S, Elkadri A, Grossman AB. North American Society for Pediatric Gastroenterology, Hepatology, and Nutrition Position Paper on the Evaluation and Management for Patients With Very Early-onset Inflammatory Bowel Disease. J Pediatr Gastroenterol Nutr. 2020 Mar;70(3):389-403. doi: 10.1097/MPG.0000000000002567. PMID 32079889
- [Result] Turner D, Otley AR, Mack D, Hyams J, de Bruijne J, Uusoue K, Walters TD, Zachos M, Mamula P, Beaton DE, Steinhart AH, Griffiths AM. Development, validation, and evaluation of a pediatric ulcerative colitis activity index: a prospective multicenter study. Gastroenterology. 2007 Aug;133(2):423-32. doi: 10.1053/j.gastro.2007.05.029. Epub 2007 May 21. PMID 17681163
- [Result] Otley A, Smith C, Nicholas D, Munk M, Avolio J, Sherman PM, Griffiths AM. The IMPACT questionnaire: a valid measure of health-related quality of life in pediatric inflammatory bowel disease. J Pediatr Gastroenterol Nutr. 2002 Oct;35(4):557-63. doi: 10.1097/00005176-200210000-00018. PMID 12394384
- [Result] Marcovitch L, Nissan A, Mack D, Otley A, Hussey S, Mclean B, Lewis M, Croft N, Barakat FM, Griffiths AM, Turner D. Item Generation and Reduction Toward Developing a Patient-reported Outcome for Pediatric Ulcerative Colitis (TUMMY-UC). J Pediatr Gastroenterol Nutr. 2017 Mar;64(3):373-377. doi: 10.1097/MPG.0000000000001259. PMID 27159210
- [Result] Taylor SJ, Whincup PH, Hindmarsh PC, Lampe F, Odoki K, Cook DG. Performance of a new pubertal self-assessment questionnaire: a preliminary study. Paediatr Perinat Epidemiol. 2001 Jan;15(1):88-94. doi: 10.1046/j.1365-3016.2001.00317.x. PMID 11237120
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921210